CLINICAL TRIAL: NCT06009367
Title: The Effect of Fascial Manipulation Technique by Stecco on the Shoulder Range of Motion and External Rotation Strength of Asymptomatic Handball Players
Brief Title: Fascial Manipulation Effect on Shoulder Range of Motion and Strength in Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anja Baric (Other)
Responsible Party: Sponsor-Investigator, Anja Baric, Principal Investigator, Physiotherapist, Master of Health Science, Anja Barič
Organization: Anja Barič (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FM2223
Record Dates: First submitted 2023-08-09; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Connective Tissue Defect; Fascia; Anomaly
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: One investigated group with intervention and one control group without intervention
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigated group with fascial manipulation (Experimental): Participants in this group received one treatment of fascial manipulation by Stecco method
  Interventions: Procedure: Fascial Manipulation by Stecco method
- Control group with no intervention (No Intervention): Participants in this group received no treatment

INTERVENTIONS:
Procedure: Fascial Manipulation by Stecco method — Fascial Manipulation (FM) is a method carefully developed by members of the Stecco family after many years of research. FM involves deep kneading of the muscle fascia at specific points called centers of coordination (CC) and centers of fusion (CF) along myofascial sequences, diagonals, and spirals. It has been proposed that the friction caused by manipulation creates localized heat and that, due to the thermosensitive characteristics of fascia, this heat facilitates the transition of hyaluronic acid within the extracellular matrix from a condensed state to a more fluid state, thus restoring the gliding properties of fascia.
  Arms: Investigated group with fascial manipulation

SUMMARY:
The investigators conducted a prospective randomized controlled trial on the female and male handball players from the Izola Handball Club (Slovenia) who volunteered to participate in the study. Data were collected in the first part of the competition season 2022/2023. The participants were randomly divided into investigated and control groups so that each group had approximately the same number of participants regarding sex and age. The Fascial manipulation (FM) was performed in the investigated group, whereas, in the control group, the participants did not receive the FM. Demographics (sex, age, height, weight, throwing shoulder, playing position, years of playing) were collected. The study protocol complied with the Declaration of Helsinki and was approved by the National Medical Ethics Committee of the Republic of Slovenia (0120-78/2022/9).

The aim of this research was to determine whether and how FM affects IR, HADD ROM and the strength of ER in handball players. The hypotheses include: (1) an increase in IR, HADD ROM, and strength of ER immediately after FM compared to the control group, (2) maintenance of increased ROM and ER strength one month after FM compared to baseline and the control group, (3) a decrease in the subjective feeling of tightness immediately and one month after and (4) the size of the FM effect increases with years of playing and vice versa.

DETAILED DESCRIPTION:
All participants aged 18 or older signed informed consent to participate in the study. For participants under 18 years of age, informed consent was signed by their parents or legal guardians. Exclusion criteria were prior upper extremity injury or upper extremity surgery preventing the player from playing in the last three months, any previous shoulder surgery, and goalkeeper position. A cluster random sampling strategy was used. The participants were randomly divided into investigated and control groups so that each group had approximately the same number of units regarding sex and age. In the investigated group, the Fascial manipulation (FM) was performed, whereas, in the control group, the participants did not receive the FM.

One session of Fascial Manipulation® by Stecco was chosen as the therapeutic procedure. The principal investigator who performed the FM in the investigated group is a qualified therapist with extensive knowledge in manual therapy and a certificate in FM Levels I and II. Based on the collected information (a complete medical history, including the chronology of any traumatic events, fractures, significant musculoskeletal dysfunctions, scars and surgical procedures, specific range of motion, and palpation examinations) and according to the Stecco model for the interpretation of the dysfunction of the fascial system, the therapist selected an individual combination of condensed points of treatment (centers of coordination - CC and/or centers of fusion - CF). All CC and/or CF points that were treated in an individual subject were recorded.

All participants completed three test sessions (pre-test, immediate post-test, and one-month post-test). The immediate post-test measurements were recorded directly after the application of the FM in the investigated group and after a one-minute waiting period in the control group. Testing was repeated 27-34 days (one month) after FM was performed. All three measurements for both groups were performed in the same way. All the measurements were performed by the two independent examiners - experienced physical therapists, whereby FM was performed only by the principal investigator-experienced physical therapist who did not participate in the measurements. Before the measurements, participants completed a specific standard warm-up for their team consisting of gentle jogging, static and dynamic full-body stretching. The warm-up was not standardized for this study.

Range of motion (ROM) measurements for internal rotation (IR) and horizontal adduction (HADD) were recorded using a classic goniometer. For the HADD assessment, participants were positioned supine on a standard examination table with both shoulders aligned. The examiner stood on top of the table, facing the participant's head, and stabilized the lateral edge of the scapula. The participant's upper limb was positioned at 90 degrees of GH abduction with 90 degrees of elbow flexion. The examiner held the subject's arm distal to the elbow and passively moved it into HADD. At the first point of resistance, a second examiner used a digital inclinometer to record the amount of motion in degrees (°) by aligning it with the humerus.

Passive IR measurements were taken with the participant lying supine on an examination table, with the shoulder at 90 degrees of abduction in the frontal plane and the elbow at 90 degrees of flexion. The examiner applied a posterior stabilizing force to the acromial process of the scapula and internally rotated the upper limb until the first point of resistance. A second investigator then recorded the amount of movement in degrees by aligning the digital inclinometer with the axis of the forearm.

The Easy Force© digital dynamometer was used to determine the strength of the external rotation (ER). Maximal isometric strength was measured in Newtons per kilogram (N/kg). Subjects lay prone, with the shoulder abducted to 90° in the frontal plane and in neutral rotation. The first examiner placed the dynamometer strap around the wrist, 2cm proximal to the ulnar styloid process. The tape on the other side of the dynamometer was fixed in a stand next to the table, in extension with the wrist. The second examiner fixed the humerus on the distal side just above the elbow to limit the motion of the humerus. According to standardized testing instructions, the procedure was as follows: one familiarization trial, then three maximal isometric tests. Participants were asked to gradually build up their strength to maximal effort over a two-second period and finally to hold their maximal effort for three seconds. The best measurement from three trials, expressed in N/kg, was used for analysis.

One session of Fascial Manipulation® by Stecco was chosen as the therapeutic procedure for the investigated group. The principal investigator who performed the FM is a qualified therapist with extensive knowledge in manual therapy and holds certificates in FM Levels I and II. The therapist utilized the Stecco model to interpret the dysfunction of the fascial system based on comprehensive information collected, including the participant's complete medical history, traumatic events, fractures, musculoskeletal dysfunctions, scars, surgical procedures, specific range of motion, and palpation examinations. Using this information, the therapist selected an individualized combination of condensed treatment points, known as centers of coordination (CC) and/or centers of fusion (CF). All CC and/or CF points treated in each individual subject were recorded for documentation purposes.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic and healthy handball players from Izola Handball Club (Slovenia)
* Both male and female participants who volunteer for the study and belong to cadet, junior, and senior handball teams
* All participants aged 18 years and older, provided informed consent to participate in the study, whereas participants under the age of 18 need their parents or guardians to sign the informed consent form on their behalf.

Exclusion Criteria:

* A recent upper extremity injury or surgery that hinders the player's ability to participate in the game of handball for the past three months
* Any history of previous shoulder surgery
* The playing position of goalkeeper.

Ages: 15 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The immediate effect of Fascial Manipulation (FM) on the shoulder joint internal rotation (IR) and horizontal adduction (HADD) range of motion (ROM) | immediately after FM
  Investigated the difference in the shoulder joint internal rotation (IR) and shoulder joint horizontal adduction (HADD) ROM before and immediately after FM in both groups. A classic goniometer was used to record ROM measurements for IR and HADD in degrees (°).
The immediate effect of Fascial Manipulation (FM) on the shoulder joint external rotation (ER) strength | immediately after FM
  Investigated the difference in the strength of ER before and immediately after FM in both groups. The Easy Force© digital dynamometer was used to determine the strength of the ER. Maximal isometric strength was measured in newtons per kilogram (N/kg).

SECONDARY OUTCOMES:
The effect of Fascial Manipulation (FM) on the shoulder joint internal rotation (IR) and horizontal adduction (HADD) range of motion (ROM) one month after FM | 27-34 days (one month)
  Investigated the difference in values of internal rotation (IR) and horizontal adduction (HADD) range of motion (ROM) one month after FM in both groups. A classic goniometer was used to record ROM measurements for IR and HADD in degrees (°).
The effect of Fascial Manipulation (FM) on the shoulder joint external rotation (ER) strength one month after FM | 27-34 days (one month)
  Investigated the difference in values of ER strength one month after FM in both groups. The Easy Force© digital dynamometer was used to determine the strength of the ER. Maximal isometric strength was measured in newtons per kilogram (N/kg).

CONTACTS AND LOCATIONS:
Locations (1):
- Izola Handball Club, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baric A, Jesensek Papez B, Bastic M, Kelc R, Brumat P, Stecco A. The Impact of Fascial Manipulation(R) on Posterior Shoulder Tightness in Asymptomatic Handball Players: A Randomized Controlled Trial. Diagnostics (Basel). 2024 Sep 7;14(17):1982. doi: 10.3390/diagnostics14171982. PMID 39272766